CLINICAL TRIAL: NCT04319835
Title: Local Metabolism of the Gastric Tube Reconstruction After Esophagectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Senzime AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U-1506
Record Dates: First submitted 2016-03-30; First posted 2020-03-24 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Microdialysis; Ischemia; Anastomotic Leakage
MeSH Terms: conditions — Ischemia; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microdialysis catheter (Experimental): Surface Microdialysis catheter will be placed onto the surgical reconstruction after esophagectomy and will be evaluated for clinical safety and performance. The metabolic profile as measured by Microdialysis will be correlated to the clinical outcome. No interventions based on the results will be performed.
  Interventions: Device: OnZurf Probe

INTERVENTIONS:
Device: OnZurf Probe

SUMMARY:
Postoperative surveillance of local metabolism of the surgical reconstruction after esophagectomy by means of Microdialysis. Dialysate is collected continuously for seven postoperative Days. Results analysed in a blinded fashion and related to the clinical outcome. Primary endpoint: anastomotic leakage

DETAILED DESCRIPTION:
The purpose of the study is to evaluate Onzurf probe (microdialysis probe) as a monitoring method for the early diagnosis of complications after surgery in the gastrointestinal tract. Samples taken with Onzurf probe will be analyzed and then compared with routine clinical data on surgical procedures in gastrointesinala tract. These parameters are: Patient general condition, endoscopy, radiology and routine clinical samples (global) as CRP (C-reactive protein), white blood cells, blood gases.The patients are their own controls when the purpose is to see if you can detect early complications with Onzurf probe and also identify how many people gets complications after surgery in the gastrointestinal tract. The patients' clinical routine tests (blood tests, etc.) will serve as control samples, which then will be compared with results from sampling of Onzurf probe. No interventions will be carried out on the patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients accepted for esophagectomy with Gastric Tube reconstruction in the Department

Exclusion Criteria:

* Surgical recontruction other than Gastric Tube

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Concentration of lactate measured by microdialysis in patients with anastomotic leakage as defined by endoscopy or radiology | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of lactate measured repeatedly (see below) to produce a metabolic profile over time
Concentration of lactate measured by microdialysis in patients with a normal uncomplicated postoperative recovery | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of lactate measured repeatedly (see below) to produce a metabolic profile over time
Concentration of glucose measured by microdialysis in patients with anastomotic leakage as defined by endoscopy or radiology | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of glucose measured repeatedly (see below) to produce a metabolic profile over time
Concentration of glucose measured by microdialysis in patients with a normal uncomplicated postoperative recovery | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of glucose measured repeatedly (see below) to produce a metabolic profile over time
Concentration of pyruvate measured by microdialysis in patients with anastomotic leakage as defined by endoscopy or radiology | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of pyruvate measured repeatedly (see below) to produce a metabolic profile over time
Concentration of pyruvate measured by microdialysis in patients with a normal uncomplicated postoperative recovery | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of pyruvate measured repeatedly (see below) to produce a metabolic profile over time
Concentration of glycerol measured by microdialysis in patients with anastomotic leakage as defined by endoscopy or radiology | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of glycerol measured repeatedly (see below) to produce a metabolic profile over time
Concentration of glycerol measured by microdialysis in patients with a normal uncomplicated postoperative recovery | Measured with four hour intervals during the first seven postoperative days
  Concentration in millimoles / liter of glycerol measured repeatedly (see below) to produce a metabolic profile over time

CONTACTS AND LOCATIONS:
Overall Officials: Jan Johansson, PhD, Principal Investigator — Region Skane
Locations (1):
- Skånes Universitetssjukhuset, Lund, Skåne County, Sweden